CLINICAL TRIAL: NCT03105427
Title: Assoziationen Von Leukozyten-Sub-Populationen im Blut kardiovaskulärer Risikopatienten Mit Der Inzidenz Perioperativer kardiovaskulärer Ereignisse
Brief Title: Leukocytes and Cardiovascular Perioperative Events-2
Acronym: LeukoCAPE-2
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Johann Motsch, Prof. Dr. med. habil., University Hospital Heidelberg
Other Study IDs: LeukoCAPE02
Record Dates: First submitted 2017-03-08; First posted 2017-04-10 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Elective Non-cardiac Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The potential use of regulatory T cells as preoperative risk stratification tool is evaluated in order to improve clinical risk stratification and reduce perioperative morbidity and mortality.

DETAILED DESCRIPTION:
Annually, there are more than 200 million surgeries worldwide. The POISE study revealed 5% of patients undergoing a non-cardiac surgery suffer perioperative myocardial infarcts going along with a perioperative mortality rate of about 11,6%. Possibilities to preoperatively identify patients at risk are limited and prophylactic interventions are not yet established or controversial.

Selected leukocyte subpopulations have been demonstrated to be associated with higher risk for cardiovascular events.

The aim of this study is to evaluate the potential use of regulatory T cells as preoperative risk stratification tool in order to improve clinical risk stratification and reduce perioperative morbidity and mortality. Therefore, high-risk cardiovascular patients scheduled for major non-cardiac surgery will be recruited. Blood will be drawn at predefined time points before surgery and up to three days postoperatively. Leukocytes will be analyzed by flow cytometry. During 30 day follow up adverse cardiovascular events will be recorded. ECGs will be recorded preoperatively and on post-OP day 3. High-sensitive cardiac Troponin T will be measured prior to the operation and on post-OP day one to three. The patient chart will be screened for cardiovascular events up to day 30. A telephone interview will be performed to detect cardiovascular events after discharge until post-OP day 30.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Coronary heart disease
* Non-cardiac surgery
* Inpatient treatment
* Informed consent

Exclusion Criteria:

* 17 years of age or younger
* Known pregnancy or breastfeeding
* Missing informed consent
* Ambulatory or day-case surgery
* Emergency surgery
* Acute or chronic leukemia
* Current aplasia or leukopenia
* Current GM-CSF treatment
* Carotid artery surgery
* History of splenectomy
* Current intravenous or oral Cortisone treatment
* History of organ transplantation
* Current immunosuppressive medication
* Chemotherapy completed less than 14 days ago
* Entity which is part of the composite endpoint diagnosed within past 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to University Hospital Heidelberg suffering coronary heart disease and scheduled for major non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Events | 30 days postoperative
  Number of participants with Cardiovascular Events defined as occurrence of Cardiac Death and/or Myocardial Ischemia and/or Myocardial Infarction and/or Myocardial Injury After Non-cardiac Surgery (MINS) and/or Embolic Stroke and/or Thrombotic Stroke recorded until postoperative day 30. Definitions according to European Perioperative Clinical Outcome-(EPCO) definitions detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days

SECONDARY OUTCOMES:
Peripheral vascular occlusion | 30 days postoperative
  Diagnosed by a radiologist based on the results of duplex ultrasonography, angiography or CT-angiography.
New onset atrial fibrillation | 30 days postoperative
  Number of participants with new electrocardiographic detection of atrial fibrillation in postoperative ECG and/or documented in patient charts
Acute kidney injury | 30 days postoperative
  Number of participants with acute kidney injury according to KDIGO guidelines
Congestive heart failure | 30 days postoperative
  Number of participants with congestive heart failure according to European Perioperative Clinical Outcome (EPCO) definitions
Cardiac death | 30 days postoperative
  Number of participants with cardiac Death defined as death because of new myocardial infarction or ischemia, or atrial or ventricular arrhythmias, or cardiogenic pulmonary edema, or pulmonary embolism detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days
Myocardial Ischemia | 30 days postoperative
  Number of participants with myocardial ischemia defined as new electrocardiographic detection of myocardial ischemia in ECG and/or documented in patient charts which will be screened up to 30 postoperative days and/or detected during telephone interview after 30 postoperative days
Myocardial Infarction | 30 days postoperative
  Number of participants with Myocardial Infarction defined as an increase in serum cardiac biomarker values in combination with symptoms of ischemia or new/presumed new significant ST segment or T wave ECG changes or new left bundle branch block or development of pathological Q waves on ECG. Definition according to European Perioperative Clinical Outcome-(EPCO) definitions detected at postoperative visits, postoperative blood analyses, documented in patient chart or detected during telephone interview after 30 postoperative days
Myocardial Injury after Non-cardiac Surgery (MINS) | 30 days postoperative
  Number of participants with MINS defined as raise in postoperative hs-cTNT (high sensitivity cardiac troponin T) jugded due to myocardial ischemia detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days
Stroke | 30 days postoperative
  Number of participants with embolic or thrombotic stroke defined cerebral event with persistent residual motor, sensory or cognitive dysfunction detected at postoperative visits, documented in patient chart or detected during telephone interview after 30 postoperative days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogacev KS, Cremers B, Zawada AM, Seiler S, Binder N, Ege P, Grosse-Dunker G, Heisel I, Hornof F, Jeken J, Rebling NM, Ulrich C, Scheller B, Bohm M, Fliser D, Heine GH. CD14++CD16+ monocytes independently predict cardiovascular events: a cohort study of 951 patients referred for elective coronary angiography. J Am Coll Cardiol. 2012 Oct 16;60(16):1512-20. doi: 10.1016/j.jacc.2012.07.019. Epub 2012 Sep 19. PMID 22999728
- [Background] Berg KE, Ljungcrantz I, Andersson L, Bryngelsson C, Hedblad B, Fredrikson GN, Nilsson J, Bjorkbacka H. Elevated CD14++CD16- monocytes predict cardiovascular events. Circ Cardiovasc Genet. 2012 Feb 1;5(1):122-31. doi: 10.1161/CIRCGENETICS.111.960385. Epub 2012 Jan 11. PMID 22238190
- [Background] Devereaux PJ, Xavier D, Pogue J, Guyatt G, Sigamani A, Garutti I, Leslie K, Rao-Melacini P, Chrolavicius S, Yang H, Macdonald C, Avezum A, Lanthier L, Hu W, Yusuf S; POISE (PeriOperative ISchemic Evaluation) Investigators. Characteristics and short-term prognosis of perioperative myocardial infarction in patients undergoing noncardiac surgery: a cohort study. Ann Intern Med. 2011 Apr 19;154(8):523-8. doi: 10.7326/0003-4819-154-8-201104190-00003. PMID 21502650
- [Background] Devereaux PJ, Sessler DI. Cardiac Complications in Patients Undergoing Major Noncardiac Surgery. N Engl J Med. 2015 Dec 3;373(23):2258-69. doi: 10.1056/NEJMra1502824. No abstract available. PMID 26630144
- [Background] Engelbertsen D, Andersson L, Ljungcrantz I, Wigren M, Hedblad B, Nilsson J, Bjorkbacka H. T-helper 2 immunity is associated with reduced risk of myocardial infarction and stroke. Arterioscler Thromb Vasc Biol. 2013 Mar;33(3):637-44. doi: 10.1161/ATVBAHA.112.300871. Epub 2013 Jan 10. PMID 23307873
- [Background] Gillmann HJ, Meinders A, Grohennig A, Larmann J, Bunte C, Calmer S, Sahlmann B, Rustum S, Aper T, Lichtinghagen R, Koch A, Teebken OE, Theilmeier G. Perioperative levels and changes of high-sensitivity troponin T are associated with cardiovascular events in vascular surgery patients. Crit Care Med. 2014 Jun;42(6):1498-506. doi: 10.1097/CCM.0000000000000249. PMID 24584063
- [Background] Kotfis K, Biernawska J, Zegan-Baranska M, Zukowski M. Peripheral Blood Lymphocyte Subsets (CD4+, CD8+ T Cells, NK Cells) in Patients with Cardiovascular and Neurological Complications after Carotid Endarterectomy. Int J Mol Sci. 2015 May 4;16(5):10077-94. doi: 10.3390/ijms160510077. PMID 25946343
- [Background] Rogacev KS, Seiler S, Zawada AM, Reichart B, Herath E, Roth D, Ulrich C, Fliser D, Heine GH. CD14++CD16+ monocytes and cardiovascular outcome in patients with chronic kidney disease. Eur Heart J. 2011 Jan;32(1):84-92. doi: 10.1093/eurheartj/ehq371. Epub 2010 Oct 12. PMID 20943670
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Size and distribution of the global volume of surgery in 2012. Bull World Health Organ. 2016 Mar 1;94(3):201-209F. doi: 10.2471/BLT.15.159293. PMID 26966331
- [Derived] Handke J, Scholz AS, Dehne S, Krisam J, Gillmann HJ, Janssen H, Arens C, Espeter F, Uhle F, Motsch J, Weigand MA, Larmann J. Presepsin for pre-operative prediction of major adverse cardiovascular events in coronary heart disease patients undergoing noncardiac surgery: Post hoc analysis of the Leukocytes and Cardiovascular Peri-operative Events-2 (LeukoCAPE-2) Study. Eur J Anaesthesiol. 2020 Oct;37(10):908-919. doi: 10.1097/EJA.0000000000001243. PMID 32516228